CLINICAL TRIAL: NCT07141082
Title: A Pilot Randomized Controlled Trial Exploring the Use of Supervised Group Art Therapy Among Older Adults With Chronic Low Back Pain: Feasibility, Potential Efficacy, and Participant Experiences
Brief Title: Expressive Art Therapy for Elder Adults With Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Prof. Fadi AL ZOUBI, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20250416004-01; 1-WZBS (Other Grant/Funding Number: Faculty Collaborative Research Scheme between Social Sciences and Health Sciences, The Hong Kong Polytechnic University)
Record Dates: First submitted 2025-08-06; First posted 2025-08-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low Back Pain
Keywords: art therapy; expressive art; chronic low back pain; Musculoskeletal Diseases; physiotherapy practice; Physical therapists; Physiotherapists
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized using cluster randomization, allocating them into two groups: the expressive art therapy plus exercises group or the exercise-only group. A research assistant not involved in the study will manage allocation. Randomization will stratify participants based on sex and functional level to ensure balanced representation in both groups.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Expressive art therapy (Experimental): One hour of expressive art therapy followed by exercise session.
  Interventions: Other: Exercise
- Control Group: Exercise (Active Comparator): The control group will be a one-hour session that includes progressive back strengthening and general reconditioning exercises, complemented by education on back care to support self-management of low back pain.
  Interventions: Other: Art therapy combined with Exercise

INTERVENTIONS:
Other: Art therapy combined with Exercise — The intervention program consists of one hour of expressive art intervention followed by one hour of exercise training. Art therapy sessions will be conducted in small groups of eight participants, facilitated by a part-time registered expressive art therapist. Each session begins with a 5-minute introduction and check-in, welcoming participants and encouraging them to share their current status. This is followed by a 10-minute mindfulness exercise designed to center participants and promote relaxation, preparing them for the creative activities ahead. The core of each session features a 20-minute art-making process focused on specific themes that guide participants in exploring their pain and personal narratives.
  Arms: Control Group: Exercise
Other: Exercise — each one-hour session in the exercise control group will involve progressive back and general reconditioning exercises, along with back care education to support self-management of LBP.
  Arms: Experimental: Expressive art therapy

SUMMARY:
This research project aims to assess the feasibility of expressive art therapy for elderly adults with chronic low back pain and to evaluate the preliminary efficacy of combining art therapy with exercise intervention. Additionally, the study will investigate facilitators and barriers to participation.

A mixed-methods approach will be employed, including a quantitative questionnaire and qualitative semi-structured focus group discussions. The questionnaire will examine physical, functional, and psychological changes potentially influenced by art therapy, while the focus groups will provide in-depth insights into participants' experiences and perceptions of the combined intervention.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is a common and debilitating condition that affects millions of older adults worldwide, significantly impacting their physical, emotional, and social well-being. This pilot randomized controlled trial (RCT) aims to explore the feasibility and potential effectiveness of a new approach that combines supervised group expressive art therapy with exercise for elderly individuals suffering from CLBP.

The primary goal is to assess participant recruitment, retention, and adherence to intervention. The investigators will also identify any logistical challenges that may arise during the process. To gather preliminary data on the intervention's effectiveness, the investigators will measure changes in pain intensity, functional ability, psychological flexibility, and health-related quality of life (HRQoL).

In addition to quantitative measures, the investigators will conduct qualitative interviews and focus groups to gain deeper insights into the participants' experiences. This will help to identify factors that facilitate or hinder their engagement with the program.

By incorporating expressive art therapy-an approach that encourages emotional expression and coping strategies-this study aims to provide a holistic method for managing pain. The ultimate goal is to enhance the quality of life for older adults affected by CLBP. If successful, this pilot RCT will offer valuable insights that could inform a larger, definitive RCT, paving the way for innovative, interdisciplinary strategies in chronic pain management and improving health outcomes in the community.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years and above
* currently experiencing non-specific low back pain for at least three months
* who have sought medical treatment for CLBP
* can read and write in Traditional Chinese
* MoCA-5 of 18 or above

Exclusion Criteria:

* malignant pain
* lumbar spinal stenosis
* confirmed dementia
* severe cognitive impairment
* serious major medical or psychiatric disorders
* currently receiving physiotherapy, cognitive therapy, or psychological treatments

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-02 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  The proportion of eligible participants who agree to enrol in the study.
Retention Rate of participants | Through study completion, an average of 8 weeks
  The proportion of participants who complete the full study protocol.
Proportion of Participants Adhering to Intervention | Weekly from week 1 through 8
  Intervention adherence will be assessed by the proportion of participants who attended at least 80% of the scheduled group sessions out of the total number randomized. Reasons for non-adherence will be explored through qualitative interviews with participants who did not meet the attendance threshold or discontinued the program prematurely.
Acceptability of the Intervention-satisfaction | Weekly from week 1 through 8
  Participants will rate their satisfaction with the program on a scale from 0 (not satisfied) to 10 (very satisfied).
Acceptability of the Intervention-perceived burden | Weekly from week 1 through 8
  Participants will rate the perceived burden of the intervention on a scale from 0 (not demanding) to 10 (very demanding).
Acceptability of the Intervention-willingness to continue | Weekly from week 1 through 8
  Participants will rate their willingness to continue with the program on a scale from 0 (not willing to continue) to 10 (very willing to continue).
Feasibility of data collection procedures | At 3-month post intervention
  This outcome measure will evaluate the feasibility and acceptability of the data collection methods used in the study, including completion rates for outcome assessments.
  Feasibility Metrics:
  Completion Rates for Outcome Assessments: The number of completed assessments will be divided by the total number of scheduled assessments to calculate the completion rate.
Safety and Adverse Events of participants | Weekly from week 1 through 8
  This outcome measure will document any adverse events or safety concerns that arise during the study, including:
  Undesirable medical occurrences or problems that a participant experiences during or after the intervention, lasting more than 2 days and/or causing the participant to seek additional treatment.
  These adverse events will be categorized into:
  Serious Related Adverse Events Non-Serious Adverse Events
  Safety Metrics:
  Number and type of adverse events Proportion of participants who report serious related adverse events Proportion of participants who report non-serious adverse events

SECONDARY OUTCOMES:
Global Impression of Change scale | Immediately post-intervention and at the 3-month follow-up post-intervention
  This is a complementary measure allows patients to self-report their impression of the overall change in their condition from the beginning of a study or intervention to the current time point. This provides a global, subjective evaluation of the patient's perceived improvement or worsening of their symptoms or health status. This item has a 7-point rating, with the following response options: very much improved, much improved, minimally improved, no change, minimally worse, much worse, and very much worse.
Numeric Pain Rating Scale (NPRS) | Baseline, immediately post-intervention, and 3 month follow up post-intervention
  An 11-point scale measuring low back pain intensity, where 0 indicates no pain and 10 indicates the worst imaginable pain. Participants need to report their back pain in the current moment, in the last 24 hours and the last 3 months.
Acceptance and Action Questionnaire II (AAQ-II) | Baseline, immediately post-intervention, and 3 month follow up post-intervention
  This 7-item Chinese version measures participants' psychological flexibility, rated on a 7-point scale, where higher scores indicate less flexibility.
  AAQ-II has been cross-culturally adapted and validated among local adolescents and has demonstrated satisfactory internal consistency and test-retest reliability
EQ-5D-5L | Baseline, immediately post-intervention, and 3 month follow up post-intervention
  The Chinese version of this instrument measures HRQoL across five domains, providing insight into participants' overall well-being.It comprises 5 items related to mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Each item has 5 response options (no problem', 'slight problems', 'moderate problems', 'severe problems', and 'extreme problems/unable to').
  It has been found to useful in monitoring treatments' effects on HRQoL.
Roland Morris Disability Index (RMDQ) | Baseline, immediately post-intervention, and 3 month follow up post-intervention
  The 24-item Chinese version of the Roland-Morris Disability Questionnaire assesses disability related to low back pain (LBP) in individuals with chronic low back pain (CLBP). Scores range from 0 to 24, with higher scores indicating greater functional limitation and worse disability.
Depression, Anxiety, and Stress Scales (DASS) | Baseline, immediately post-intervention, and 3 month follow up post-intervention
  The 21-item Chinese version evaluates mental health across three domains, with higher scores indicating greater issues. It has been cross-culturally adapted to Hong Kong settings,demonstrating excellent internal consistency for depression, anxiety, and stress subscales.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Sciences, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
All personal data will be anonymized. The investigators will minimize the use of personal data in the study as much as possible. The data will be kept for 5 years after project completion, with limited access by Dr. Fadi Al Zoubi.